CLINICAL TRIAL: NCT06075550
Title: Assessment of Postoperative Pain of Two Bioceramic Root Canal Sealers After Different Obturation Techniques: A Randomized Clinical Trial
Brief Title: Assessment of Postoperative Pain of Two Bioceramic Root Canal Sealers With Obturation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hussein Amr Youssef Shoukry, Phd student-endodontic department, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 439
Record Dates: First submitted 2023-04-21; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Effect of Material and Technique

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TotalFill BC Sealer (Experimental): single cone technique with TotalFill BC Sealer
  Interventions: Other: single cone technique using TotalFill BC Sealer; Other: warm vertical compaction technique using TotalFill BC Sealer HiFlow
- TotalFill BC Sealer HiFlow (Experimental): warm vertical compaction technique with TotalFill BC Sealer HiFlow
  Interventions: Other: single cone technique using TotalFill BC Sealer; Other: warm vertical compaction technique using TotalFill BC Sealer HiFlow

INTERVENTIONS:
Other: single cone technique using TotalFill BC Sealer — Gutta percha cone size X5 (Dentsply, Maillefer) TotalFill BC Sealer (FKG Dentaire SA, La Chaux-de-Fonds, Switzerland)
Other: warm vertical compaction technique using TotalFill BC Sealer HiFlow — TotalFill BC Sealer HiFlow (FKG Dentaire SA, La Chaux-de-Fonds, Switzerland)

SUMMARY:
60 patients were divided into 2 groups, 30 patient in each group

Group I: Obturation with TotalFill BC Sealer using the single cone technique

Group II: Obturation with TotalFill BC Sealer HiFlow using the warm vertical compaction technique.

Every participant will be given a Visual Analog Scale (VAS) to record the intensity of postoperative pain at 6 hr, 24 hr, 48 hr, 72 hr, and 1week after treatment. The patients will return their Visual Analog Scale (VAS) after 1 week and the recorded pain data will be collected and statistically analyzed regarding each group.

DETAILED DESCRIPTION:
Endodontic treatment will be performed in a single visit

Root canal preparation

* After anesthesia a rubber dam will be placed then disinfection of the working field will be done using sodium hypochlorite swab.
* All caries will be removed then an endodontic access cavity will be established using high speed carbide burs under coolant.
* Cleaning and shaping of the canal will be performed using rotary ProTaper Next files (Dentsply, Maillefer) connected to an endodontic motor according to the manufacturer's instructions and recommendations.
* Irrigation with sodium hypochlorite will be always performed during instrumentation.
* After instrumentation a final flush with sodium hypochlorite followed by distilled water will be performed and the canals will be dried using sterile paper points.
* Master cone radiograph will be taken for confirmation and obturation will be done according to the mentioned groups.

Root canal obturation

* This study will be a double blind randomized study.
* Group I: Using TotalFill BC Sealer, the tip of the syringe will be inserted into the canal and the sealer will be dispensed into the root canal as recommended by the manufacturer. A ProTaper Next gutta percha cone (Dentsply, Maillefer) of the same size of the prepared canal will be used for single cone obturation technique and the excess gutta percha will be removed by a heated condenser.
* Group II: TotalFill BC Sealer HiFlow will be inserted into the canal as in Group I and the master gutta percha cone will be placed and warm vertical compaction technique will be done. The depth of the heated plugger will be 5 mm less than the WL followed by back filling.
* After obturation, the access cavity will be cleaned and a sterile cotton pellet is placed and the cavity will be sealed with temporary filling.
* A postoperative radiograph will be taken

Assessment of postoperative pain

Every participant will be given a Visual Analog Scale (VAS) to record the intensity of postoperative pain at 6 hr, 24 hr, 48 hr, 72 hr, and 1week after treatment. The patients will return their Visual Analog Scale (VAS) after 1 week and the recorded pain data will be collected and statistically analyzed regarding each group.

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients
* Patients age between 20-50 years
* Vital pulp as indicated by thermal or electric pulp test
* No history of previously initiated root canal treatment among the treated tooth
* Sufficient tooth structure for isolation
* Teeth with mature apices

Exclusion Criteria:

* Pregnancy or lactation
* Medically compromised patients
* Previous endodontic therapy of the tooth to be treated.
* Teeth diagnosed with non-vital pulp.
* Periodontally compromised teeth (teeth with periodontal probing depth more than 3mm).
* Teeth with abnormal anatomy or calcified canals.
* Teeth with caries below the bony level (non-restorable tooth).
* Immature teeth with open apices.
* Complications during treatment (file separation, ledges, perforation, etc.)
* Overfilling (overextended beyond the radiographic apex) or short filling (more than 2mm of the radiographic apex)
* Radiographic evidence of root resorption
* Patients who could not follow the instructions to record the visual analog scale

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
change of postoperative pain (Visual Analog Scale ) | postoperative pain at 6 hours
  numerical (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and dental medicine, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Result] Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011 Apr;37(4):429-38. doi: 10.1016/j.joen.2010.12.016. PMID 21419285
- [Result] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J. 2008 Feb;41(2):91-9. doi: 10.1111/j.1365-2591.2007.01316.x. Epub 2007 Oct 23. PMID 17956561
- [Result] El Mubarak AH, Abu-bakr NH, Ibrahim YE. Postoperative pain in multiple-visit and single-visit root canal treatment. J Endod. 2010 Jan;36(1):36-9. doi: 10.1016/j.joen.2009.09.003. PMID 20003932